CLINICAL TRIAL: NCT05199181
Title: An Approach Feasibility Study to Establish Full Pulpotomy in Mature Teeth With Symptomatic Irreversible Pulpitis as a Routine Treatment in the Primary Care Dental Clinics of the Public Health System in Mexico
Brief Title: Full Pulpotomy in Mature Teeth With Symptomatic Irreversible Pulpitis as a Routine Treatment in the Primary Care Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rubén Domínguez Pérez (Other)
Responsible Party: Sponsor-Investigator, Rubén Domínguez Pérez, Head of department Multidisciplinary Dentistry Research, Universidad Autónoma de Querétaro
Organization: Universidad Autónoma de Querétaro (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS1/ENS/215/220
Record Dates: First submitted 2022-01-03; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: symptomatic irreversible pulpitis; full pulpotomy; mature teeth

STUDY DESIGN:
Intervention Model Description: Longitudinal prospective single-arm cohort clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Full pulpotomy (Experimental): All patients were treated in one visit (with Full Pulpotomy); the previously trained General Practice Dentist performed all the clinical procedures
  Interventions: Procedure: Full pulpotomy

INTERVENTIONS:
Procedure: Full pulpotomy — After applying the rubber dam. Caries, and weak tissues were removed, and the endodontic access was prepared with a carbide bur. Most of the pulp was removed with a sterile high-speed diamond bur under sterile saline solution irrigation and amputated to the canal orifices level. Hemostasis was achieved by irrigation of the cavity with the same solution and an application of small cotton pellets for max.10 min. White Mineral Trioxide Aggregate was mixed according to the manufacturer´s instructions and was placed against the wound after successful hemostasis using an amalgam carrier and packed using an amalgam standard condenser. The material was adapted and a moistened cotton pellet was placed directly over the Mineral Trioxide Aggregate. After 15 minutes, the cotton was removed and the tooth was restored with amalgam. A postoperative radiograph was taken after restoration, general care instructions were given to the patients, and the recommendation of three analgesic intakes.

SUMMARY:
The present study has the objective of being a first approach of the full feasibility study in order to find out whether the Full Pulpotomy performed by a general practice dentist in a primary care dental clinic at the public health system with limited armamentarium could be suitable and present an appropriate success rate as well as patient satisfaction.

DETAILED DESCRIPTION:
The present study has the objective of being a first approach of the full feasibility study in order to find out whether the Full Pulpotomy performed by a general practice dentist in a primary care dental clinic at the public health system with limited armamentarium could be suitable and present an appropriate success rate as well as patient satisfaction. This information will help to decide if a multi-center non-randomized intervention designed study is carried out to determine if it is feasible to provide Full Pulpotomy as a routine treatment to symptomatic irreversible pulpitis or caries pulp exposure at the primary care dental clinics of the public health system in Mexico.

ELIGIBILITY:
Inclusion Criteria:

All the patients attending the primary care dental clinic with deep caries and/or pain in a permanent premolar or molar tooth.

* Teeth with complete radicular growth.
* Preoperative symptoms of irreversible pulpitis (Spontaneous pain or exacerbated by thermal stimuli and lasting for a few seconds to several hours interpreted as lingering pain compared with a control tooth and that could be reproduced using thermal testing)

Exclusion Criteria:

Medically comprised or pregnant patients.

* Teeth exclusion criteria:
* Pathological mobility
* Sinus tract
* Teeth that cannot be restored with amalgam
* Radiographic internal or external resorption
* Presence of apical rarefaction

Ages: 17 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Treatment success rate | 1 Month follow-up
  To be considered successful, none of the following symptoms had to be present at one month follow-up: persistent pain, exaggerated tenderness to percussion, pathologic mobility, swelling, sinus track related to the treated tooth, evidence of periradicular radiolucency, furcal pathosis, or root resorption
Treatment success rate | 3 Months follow-up
  To be considered successful, none of the following symptoms had to be present at three months follow-up: persistent pain, exaggerated tenderness to percussion, pathologic mobility, swelling, sinus track related to the treated tooth, evidence of periradicular radiolucency, furcal pathosis, or root resorption
Treatment success rate | 6 Months follow-up
  To be considered successful, none of the following symptoms had to be present at six months follow-up: persistent pain, exaggerated tenderness to percussion, pathologic mobility, swelling, sinus track related to the treated tooth, evidence of periradicular radiolucency, furcal pathosis, or root resorption
Treatment success rate | 9 Months follow-up
  To be considered successful, none of the following symptoms had to be present at nine months follow-up: persistent pain, exaggerated tenderness to percussion, pathologic mobility, swelling, sinus track related to the treated tooth, evidence of periradicular radiolucency, furcal pathosis, or root resorption
Treatment success rate | 12 Months follow-up
  To be considered successful, none of the following symptoms had to be present at 12 months follow-up: persistent pain, exaggerated tenderness to percussion, pathologic mobility, swelling, sinus track related to the treated tooth, evidence of periradicular radiolucency, furcal pathosis, or root resorption

SECONDARY OUTCOMES:
Satisfaction with the effect of the treatment | 24 Hours
  Patients were contacted by phone to record the satisfaction with the effect of the treatment. The possible answers for their satisfaction level were: "Very satisfied", "Satisfied", "Neither satisfied nor dissatisfied", "Dissatisfied", or "Very dissatisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Sanchez-Lara y Tajonar, DDS, Endod, Study Director — Universidad Autónoma de Querétaro
Locations (1):
- Centro de Salud -La Negreta- Jurisdicción Sanitaria 1 del Estado de Querétaro, Querétaro, Mexico